CLINICAL TRIAL: NCT01096524
Title: Phase III Study Investigating the Effects of 6-weeks of Neuromuscular Electrical Stimulation (NMES) Peri-total Knee Arthroplasty (TKA).
Brief Title: Effects of Kneehab 12-week Peri-operative Total Knee Arthroplasty
Acronym: KneehabTKA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio-Medical Research, Ltd. (Industry)
Collaborators: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BMR-09-1007; 2008-008483-27 (EudraCT Number)
Record Dates: First submitted 2010-03-24; First posted 2010-03-31 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2013-08

CONDITIONS: Knee Osteoarthritis; Disuse Atrophy
Keywords: Kneehab; NMES; Total Knee Arthroplasty; Total Knee Replacement; TKA; Disuse atrophy; muscle hypertrophy; TKR; Atrophy Prevention
MeSH Terms: conditions — Osteoarthritis, Knee; Muscular Disorders, Atrophic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group standard physiotherapy (Other): Standard pathway of care pre-and post-TKA without using NMES.
  Interventions: Other: Standard Physiotherapy
- Kneehab (Experimental): Kneehab on the quadriceps of the affected leg, 20 minutes, twice per day, 5 days per week over 12-week intervention (6 weeks pre-op, 6 weeks post op).
  Interventions: Device: Kneehab

INTERVENTIONS:
Other: Standard Physiotherapy — The Control group will complete the standard physiotherapy care pre and post-TKA surgery without NMES.
  Arms: Control group standard physiotherapy
Device: Kneehab — NMES 2 x 20 minute sessions/day, 5 days/week, 6 weeks pre and 6 weeks post TKA.
  Kneehab™ (Bio-Medical Research, Ltd., Galway, Ireland) is a NMES device with Multipath™ technology, designed to activate the quadriceps muscle. Kneehab™ is a battery operated, portable, 2-channel cutaneous electrical muscle stimulator, which operates using constant current pulses to stimulate the nerves innervating the quadriceps muscle. Kneehab™, consists of a thigh wrap with anatomically shaped electrodes and a control unit. Electrodes are placed over the quadriceps muscles and the garment is wrapped around the leg above the knee. Brief electrical impulses are delivered through the skin surface adhesive electrodes.
  Other Names: Neuromuscular Electrical Stimulation; NMES
  Arms: Kneehab

SUMMARY:
Determine the efficacy of neuromuscular electrical stimulation (NMES, Kneehab) in promoting accelerated recovery of quadriceps function in patients recovering from total knee arthroplasty (TKA) as measured by increases in isometric strength of the knee extensors and scores in the Timed Up and Go (TUG) test.

DETAILED DESCRIPTION:
Knee osteoarthritis is a severe debilitating condition that greatly impacts patient quality of life, function, emotional well-being and everyday pain levels. Total knee arthroplasty (TKA) is performed as a means of alleviating these symptoms in the long term however short term muscle weakness following surgery can elicit its own detrimental effect on performance and activities of daily living. This underlines the importance of mitigating strength loss in the immediate post-operative period.

Recent reviews suggest that Neuromuscular Electrical Stimulation (NMES) of the quadriceps femoris muscle can be beneficial in the rehabilitation period following knee surgery. It appears that early use of NMES can help to recover exercise capacity in the muscle, thus allowing the patient to benefit more from volitional exercise therapy later in the rehabilitation period1. This in turn can lead to accelerated recovery and improved outcomes. A recent and as yet unpublished study of 96 patients following ACL reconstruction has demonstrated a clear benefit to the use of Kneehab. The benefit seemed to accrue in the six-week post-operative period.

A recent pilot study by Walls 2 also suggests that NMES applied in the immediate pre-operative period before TKA leads to increased muscle strength and improved functional abilities. Previously, Mizner (2005) has shown pre operative strength to be a good predictor of functional outcome 1 year after surgery3. This proposed study aims to examine whether NMES applied in the peri-operative timeframe, 6 weeks before and 6 weeks after, can improve outcomes for patients undergoing total knee replacement. The rationale for this approach is that NMES can help prepare the quadriceps muscle for the rehabilitation phase by building exercise capacity before the operation. The immediate deficit, which normally follows knee surgery, would therefore be compensated to some extent and the post-operative NMES treatment would be expected to counteract the activation inhibition that is thought to occur in the early weeks following surgery. Overall, the patient would be in a better position to benefit from conventional rehabilitation exercises aimed at improved co-ordination and functional performance.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are scheduled for elective Total Knee Replacement surgery
* Individuals who are at least 18 years of age
* Individuals with a body mass index (BMI) <40
* Individuals who are walking independently with or without assistive devices
* Must be able and willing to complete all study assessments and to be followed for the full course of the study.
* Must be able to read, write and follow instructions in English.
* Must be able and willing to provide informed consent.
* Must be willing and able to attend for pre-op assessment

Exclusion Criteria:

* Individuals who have failed the pre-operative assessment
* Individuals with a history of foot and/or ankle pathology
* Individuals with a history of tibial or femoral fractures
* Individuals with a history of underlying neurological conditions
* Individuals with physical conditions which would make them unable to perform study procedures
* Individuals with a total hip replacement
* Individuals undergoing revision TKA of the same operated leg
* Pregnant women or inadequate precautions to prevent pregnancy
* Diagnosis of a medical condition that would contraindicate treatment with the product,e.g skin lesions at electrode site.
* Individuals with an active implanted medical device (i.e. pacemaker, pump)
* Individuals with a history of stroke
* Individuals with a history of neurological disorder that affects lower extremity function (stroke, peripheral neuropathy, Parkinson's disease, multiple sclerosis, etc.)
* Individuals with a diagnosis of inflammatory arthritis (including Rheumatoid Arthritis, gout or psoriatic arthritis)
* Individuals with muscle disease (i.e. muscular dystrophy)
* Visible skin injury or disease on their legs
* Principal investigator for this study, or member of study staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of Kneehab in promoting early recovery of quadriceps performance following knee arthoplasty. | 6 weeks Pre-Op and 6, 12 and 52 weeks post op.
  Isometric muscle strength of the knee extensors will be measured by dynamometer with the knee flexed to 60°.
  Functional ability will be measured using the Timed Get Up and Go (TUG) and Stair Climb Test (SCT).

SECONDARY OUTCOMES:
Determine the effect of Kneehab in promoting quality of life measures and health economic outcomes, compared to controls. | 6 Weeks pre-Op and 6, 12 and 52 weeks post-Op
  Administration of the Western Ontario McMaster University Osteoarthritis Index (WOMAC) and The Medical Outcomes Survey (SF-12). Health economic data will include patient length of stay post surgery; number of outpatient physiotherapy visits in the following year, and change in analgesic medication use during the 6 weeks pre- and 12 weeks post surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Alasdair Santini, M.D., Principal Investigator — Royal Liverpool & Broadgreen University Hospital
Locations (1):
- Royal Liverpool and Broadgreen University Hospital NHS Trust, Liverpool, Liverpool, United Kingdom

REFERENCES:
- [Background] Paillard T. Combined application of neuromuscular electrical stimulation and voluntary muscular contractions. Sports Med. 2008;38(2):161-77. doi: 10.2165/00007256-200838020-00005. PMID 18201117
- [Background] Mizner RL, Petterson SC, Stevens JE, Axe MJ, Snyder-Mackler L. Preoperative quadriceps strength predicts functional ability one year after total knee arthroplasty. J Rheumatol. 2005 Aug;32(8):1533-9. PMID 16078331
- [Background] Stevens JE, Mizner RL, Snyder-Mackler L. Quadriceps strength and volitional activation before and after total knee arthroplasty for osteoarthritis. J Orthop Res. 2003 Sep;21(5):775-9. doi: 10.1016/S0736-0266(03)00052-4. PMID 12919862
- [Background] Kennedy DM, Stratford PW, Hanna SE, Wessel J, Gollish JD. Modeling early recovery of physical function following hip and knee arthroplasty. BMC Musculoskelet Disord. 2006 Dec 11;7:100. doi: 10.1186/1471-2474-7-100. PMID 17156487